CLINICAL TRIAL: NCT01353040
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AVI-6003 in Healthy Adult Volunteers
Brief Title: Safety Study of Single Administration Post-exposure Prophylaxis Treatment for Marburg Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6003-us-101; W9113M-10-C-0056 (Other Grant/Funding Number: Transformational Medical Technologies, US Dept. of Defense)
Record Dates: First submitted 2011-04-22; First posted 2011-05-12 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Marburg Hemorrhagic Fever
MeSH Terms: conditions — Marburg Virus Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVI-6003 (Experimental): Phosphorodiamidate morpholino antisense oligomer with positive charges on selected subunits (PMOplus™)
  Interventions: Drug: AVI-6003
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVI-6003 — Single intravenous administration
  Arms: AVI-6003
Drug: Placebo — Single intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and pharmacology of single administrations of AVI-6003, a post-exposure prophylaxis candidate treatment for Marburg virus.

DETAILED DESCRIPTION:
Marburg hemorrhagic fever is a rare human disease caused by the Marburg virus, a filamentous, single-stranded, negative-sense RNA virus. In general, the mortality rate associated with Marburg virus outbreaks has ranged from 23% to 88%, with the highest death rates seen in more recent epidemics. No vaccine or effective therapy is available for Marburg hemorrhagic fever. AVI-6003 is an experimental combination of 2 phosphorodiamidate morpholino antisense oligomers with positive charges on selected subunits (PMOplus™). These oligomers specifically target viral messenger RNA encoding 2 Marburg virus proteins thought to be important in viral replication and host immune suppression. The present study is designed to characterize the safety, tolerability and pharmacokinetics of escalating single-administration doses of AVI-6003 in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and between the ages of 18 and 50 years in good general health
* Volunteers must be willing to use barrier methods of contraception or be of non-childbearing potential
* Volunteers must be willing to undergo a urine screen for drugs of abuse

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Any clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis
* Positive test for human immunodeficiency virus, hepatitis B or hepatitis C or known history of HIV infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events | 28 days

SECONDARY OUTCOMES:
Plasma drug concentration | 28 days
Urine drug concentration | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alison Heald, MD, Study Director — Sarepta Therapeutics, Inc.; Apinya B Vutikullird, MD, Principal Investigator — West Coast Clinical Trials
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States